CLINICAL TRIAL: NCT02621970
Title: Randomized Phase 3 Trial of Triple Combination of Induction, Concurrent and Adjuvant Chemotherapy Versus Concurrent Chemotherapy Alone in High Risk Nasopharyngeal Carcinoma Patients Treated With Intensity-modulated Radiotherapy
Brief Title: Effect of Triple Combination of Induction, Concurrent and Adjuvant Chemotherapy in High Risk Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); The First Affiliated Hospital of Guangdong Pharmaceutical University (Other)
Responsible Party: Principal Investigator, Fang-Yun Xie, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-FXY-098-Dept. of RT
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — SSRP1 protein, human; cisplatin-guanosine adduct; Docetaxel; Capecitabine; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IC plus CC plus IMRT plus AC (Experimental): Induction chemotherapy: TP -- Docetaxel 75mg/m2, D1 and cisplatin 25 mg/m2, D1-3 every 3 weeks for 2 cycles; Concurrent chemotherapy: PX -- Cisplatin 25 mg/m2, D1-3 and Xeloda 2000mg/m2, D1-14, every 3 weeks for 3 cycles; Radiation: Intensity-modulated radiotherapy; Adjuvant chemotherapy: Xeloda 2500mg/m2, D1-14, every 3 weeks for 2 cycles
  Interventions: Drug: Cisplatin 1; Drug: Docetaxel; Drug: Xeloda; Radiation: Intensity-modulated radiotherapy
- CC plus IMRT (Active Comparator): Concurrent chemotherapy: Cisplatin 100 mg/m2, D1, every 3 weeks for 3 cycles; Radiation: Intensity-modulated radiotherapy
  Interventions: Drug: Cisplatin 2; Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Cisplatin 1 — Cisplatin 25 mg/m2, D1-3
  Other Names: DDP
  Arms: IC plus CC plus IMRT plus AC
Drug: Cisplatin 2 — Cisplatin 100 mg/m2, D1
  Other Names: DDP
  Arms: CC plus IMRT
Drug: Docetaxel — Docetaxel 60mg/m2, D1
  Other Names: T
  Arms: IC plus CC plus IMRT plus AC
Drug: Xeloda — Xeloda 2000mg/m2, D1-14 in concurrent chemotherapy and Xeloda 2500mg/m2, D1-14 in adjuvant chemotherapy
  Other Names: X
  Arms: IC plus CC plus IMRT plus AC
Radiation: Intensity-modulated radiotherapy — Intensity-modulated radiotherapy
  Other Names: IMRT

SUMMARY:
The investigators aim to evaluate the survival benefit from triple combination of induction, concurrent and aduvant chemotherapy versus concurrent chemotherapy alone for high risk locoregionally advanced nasopharyngeal carcinoma treated with intensity-modulated radiotherapy.

DETAILED DESCRIPTION:
All eligible patients receive intensity-modulated radiotherapy (IMRT) with a total dose of 68 to 70 Gy in 33 fractions to the primary tumor. Patients in the experimental arm receive triple therapy of induction, concurrent and adjuvant chemotherapy. Induction chemotherapy consists of docetaxel 75 mg/m², D1 and cisplatin 25 mg/m², D1-3 every 3 weeks for 2 cycles. Concurrent chemotherapy in the experimental arm consists of cisplatin 25 mg/m², D1-3 every 3 weeks and Xeloda 2000mg/m², D1-14 for 3 cycles. Adjuvant chemotherapy consists of Xeloda 2500mg/m², D1-14 for 2 cycles. Concurrent chemotherapy in the control arm consists of cisplatin 100 mg/m², D1 every 3 weeks for 3 cycles.The primary endpoint is failure-free survival (FFS). Secondary end points include overall survival (OS), locoregional relapse-free survival (LRFS), distant metastasis-free survival (DMFS) and the incidence of grade 3 or higher acute toxicities. All efficacy analyses are conducted in the intention-to-treat population, and the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly histologically confirmed non-keratinizing (WHO 1991) nasopharyngeal carcinoma.
* Tumor staged as T4N0-3M0 or T1-3N3M0 (the 2010 UICC/AJCC staging system).
* Pretreatment EBV DNA ≥ 4000 copies/mL.
* Karnofsky scale (KPS) ≥ 70.
* Adequate marrow: leucocyte count ≥ 4×10E9/L, hemoglobin ≥ 110g/L and platelet count ≥ 100×10E9/L.
* Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and bilirubin ≤ 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤ 2.5×ULN.
* Adequate renal function: creatinine clearance ≥ 60 ml/min or creatinine ≤ 1.5×ULN.
* Patients must give written informed consent.

Exclusion Criteria:

* Prior malignancy, except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
* Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).
* History of previous radiotherapy (except for non-melanomatous skin cancers outside intended radiotherapy volume).
* Prior radiotherapy, chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance.
* Dihydropyrimidine dehydrogenase deficiency.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 534 (Estimated)
Dates: Start 2016-01; Primary Completion 2022-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
failure-free survival | Two year

SECONDARY OUTCOMES:
overall survival | two year
distant metastasis-free survival | two year
locoregional relapse-free survival | two year
Number of participants with treatment-related acute adverse events as assessed by CTCAE v4.0 | two months

CONTACTS AND LOCATIONS:
Overall Officials: Fang-Yun Xie, M.D., Principal Investigator — Sun Yat-sen University Cancer Center,Guangzhou, Guangdong, China
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hui EP, Ma BB, Leung SF, King AD, Mo F, Kam MK, Yu BK, Chiu SK, Kwan WH, Ho R, Chan I, Ahuja AT, Zee BC, Chan AT. Randomized phase II trial of concurrent cisplatin-radiotherapy with or without neoadjuvant docetaxel and cisplatin in advanced nasopharyngeal carcinoma. J Clin Oncol. 2009 Jan 10;27(2):242-9. doi: 10.1200/JCO.2008.18.1545. Epub 2008 Dec 8. PMID 19064973
- [Background] Lee AW, Ngan RK, Tung SY, Cheng A, Kwong DL, Lu TX, Chan AT, Chan LL, Yiu H, Ng WT, Wong F, Yuen KT, Yau S, Cheung FY, Chan OS, Choi H, Chappell R. Preliminary results of trial NPC-0501 evaluating the therapeutic gain by changing from concurrent-adjuvant to induction-concurrent chemoradiotherapy, changing from fluorouracil to capecitabine, and changing from conventional to accelerated radiotherapy fractionation in patients with locoregionally advanced nasopharyngeal carcinoma. Cancer. 2015 Apr 15;121(8):1328-38. doi: 10.1002/cncr.29208. Epub 2014 Dec 19. PMID 25529384
- [Background] Chen L, Hu CS, Chen XZ, Hu GQ, Cheng ZB, Sun Y, Li WX, Chen YY, Xie FY, Liang SB, Chen Y, Xu TT, Li B, Long GX, Wang SY, Zheng BM, Guo Y, Sun Y, Mao YP, Tang LL, Chen YM, Liu MZ, Ma J. Concurrent chemoradiotherapy plus adjuvant chemotherapy versus concurrent chemoradiotherapy alone in patients with locoregionally advanced nasopharyngeal carcinoma: a phase 3 multicentre randomised controlled trial. Lancet Oncol. 2012 Feb;13(2):163-71. doi: 10.1016/S1470-2045(11)70320-5. Epub 2011 Dec 7. PMID 22154591
- [Background] Wu F, Wang R, Lu H, Wei B, Feng G, Li G, Liu M, Yan H, Zhu J, Zhang Y, Hu K. Concurrent chemoradiotherapy in locoregionally advanced nasopharyngeal carcinoma: treatment outcomes of a prospective, multicentric clinical study. Radiother Oncol. 2014 Jul;112(1):106-11. doi: 10.1016/j.radonc.2014.05.005. Epub 2014 Jun 2. PMID 24933452
- [Background] Zhang LN, Gao YH, Lan XW, Tang J, OuYang PY, Xie FY. Effect of taxanes-based induction chemotherapy in locoregionally advanced nasopharyngeal carcinoma: A large scale propensity-matched study. Oral Oncol. 2015 Oct;51(10):950-6. doi: 10.1016/j.oraloncology.2015.07.004. Epub 2015 Jul 21. PMID 26209065